CLINICAL TRIAL: NCT05953090
Title: VALOR: Vaginal Atrophy & Long-term Observation of Recovery
Acronym: VALOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stratpharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPAMG03
Record Dates: First submitted 2023-03-29; First posted 2023-07-19 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Atrophic Vaginitis; Vaginal Atrophy; Genitourinary Syndrome of Menopause; Lichen Sclerosus of Vulva; Lichen Planus of Vulva; Lichen Simplex of Vulva (Disorder)
MeSH Terms: conditions — Atrophic Vaginitis; Vulvar Lichen Sclerosus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Feasibility (Experimental)
  Interventions: Device: 7-0940

INTERVENTIONS:
Device: 7-0940 — A non-hormonal and non-steroidal gel that supports vulvovaginal mucosal conditions and speeds up recovery post vaginal rejuvenation. It is a suitable alternative to vaginally administered estrogen and topical corticosteroids, that promotes a moist healing environment leading to faster re-epithelialization. The gel relieves symptoms such as itchiness, tenderness, dryness, burning sensation, painful intercourse (dyspareunia), painful urination (dysuria), rectal and defecating pain. It improves erythema, mucosal tissue thinning, erosions, fissures, ulcerations, scarring/adhesions and swelling. It is indicated for long-term use to maintain the health of the vaginal mucosa without the side effects of vaginally administered hormonal therapy and topical corticosteroids.
  Other Names: StrataMGT

SUMMARY:
Vulvovaginal skin conditions, namely vaginal atrophy, lichen sclerosus, lichen simplex chronicus and lichen planus affecting the female adult population will be treated with a novel gel dressing to test the short- and long-term safety and efficacy of the device.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed atrophic vaginitis, lichen sclerosus, lichen simplex chronicus or lichen planus
* Continuous vulvovaginal symptoms
* Access to smartphone and tablet, laptop or computer
* Access to a valid email address

Exclusion Criteria:

* Unable to provide informed consent
* Patient unable to apply topical device
* Allergy or intolerance to ingredients or excipients of the formulation of studied products
* Systemic hormonal therapy started less than 30 days before baseline
* Systemic corticosteroids ongoing treatment or used within the last 30 days before baseline
* Ongoing topical HRT or corticosteroid treatment for the indication under investigation
* Topical HRT or corticosteroid treatment used for the indication under investigation within the last 30 days before baseline

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Vulvovaginal Symptoms Questionnaire (VSQ) score from baseline at 12 months. | 12 months
  The patient-rated quality of life will be assessed at baseline and during each monthly follow-up using the validated patient-rated Vulvovaginal Symptoms Questionnaire (VSQ) [min:0; max:16 (for sexually inactive patients) / max: 20 (for sexually active patients)]. A higher score thereby correlates to a worse outcome. The primary endpoint is the change from baseline VSQ score at 12 months.
Change in Vulvar Disease Quality of Life Index (VQLI) score from baseline at 12 months | 12 months
  The patient-rated quality of life will be assessed at baseline and during each monthly follow-up using the validated patient-rated Vulvar Disease Quality of Life Index (VQLI). [min:0; max:45]. A higher score thereby correlates to a worse outcome. The primary endpoint is the change from baseline VQLI score at 12 months.

SECONDARY OUTCOMES:
Change in investigator-rated severity of visual clinical signs related to the disease, assessed using a 10-point Likert scale | 12 months
  Signs (dryness, tissue thinning, erosion, fissures, erythema, scarring, contact bleeding, labial fusion, labia reabsorption and contracture of posterior introitus) are rated by the investigator during a physical assessment at baseline and after 12 months, using a 10-point Likert scale ranging from 0=normal to 10=worst possible.
Change in patient-rated symptom severity assessed using a 10-point Likert scale. | 12 months
  Severity of symptoms (itch, burning, pain, irritation, dryness and pain during intercourse) are rated by the patient at baseline and at 12 months, using a 10-point Likert scale ranging from 0=normal to 10=worst possible.
Change in investigator-rated severity of the overall visual pathology of the disease, assessed using a 10-point Likert scale. | 12 months
  Severity of the visual pathology is rated by the investigator during baseline and after 12 months, using a 10-point Likert scale, ranging from 0=normal to 10=worst possible. Overall visual severity may include the severity of pathology at the Clitoral Hood, Urethra Area, Vaginal Vault, Labia Majora / Minora, Fourchette, Perineum, Perianal skin, Extragential site and/or Inguinal folds.
Adverse Reactions | 12 months
  Adverse reactions are rated by the investigator during baseline and after months 3, 6, 9, 12 months, using the dichotomous scale of presence and absence.
Product rating | 12 months
  Product performance is rated by the patient at the final visit after 12 months, using a Likert scale from 1=unsatisfactory to 5=excellent.
Treatment adherence | 12 months
  Treatment adherence is reported by the patient during the final study assessment, indicating the number of days/week and times/day the product was applied during the previous month. Percentage of treatment adherence is calculated from the minimum required treatment schedule.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Orange Coast Women's Medical Group, Laguna Hills, California
  - WR-PRI, LLC (Los Alamitos), Los Alamitos, California
  - WR-PRI, LLC (Newport Beach), Newport Beach, California
  - WR-Women's Health Care Research, LLC, San Diego, California
  - WR-Multi-Specialty Research Associates, Lake City, Florida
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - WR-Clinical Research Center of Nevada, LLC, Las Vegas, Nevada
  - WR-Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - WR-Charleston Clinical Trials, LLC, Charleston, South Carolina
  - Southern Urogynecology, West Columbia, South Carolina
  - WR-Medical Research Center of Memphis, LLC, Memphis, Tennessee
  - WR-Global Medical Research, LLC, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No